CLINICAL TRIAL: NCT02781935
Title: Diffusion-Weighted Magnetic Resonance Imaging Assessment of Liver Metastasis to Improve Surgical Planning
Brief Title: Diffusion-Weighted MRI for Liver Metastasis
Acronym: DREAM
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Japan Clinical Oncology Group (Other); European Society of Surgical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: EORTC-1527-GITCG-IG
Record Dates: First submitted 2016-05-17; First posted 2016-05-25 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer; Colon Cancer Liver Metastasis; Malignant Neoplasm of Rectum Metastatic to Liver
Keywords: unresectable colorectal liver metastasis; diffusion weighted MRI; disappearing liver metastasis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: DW-MRI — DW-MRI combined with Contrast Enhanced MRI will be used to confirm the status of disappearing liver metastasis prior to surgery and will be compared to findings from either histopathology of resected lesions (Rubbia-Brandt Classification of Tumor regression grading) or follow-up imaging of lesions left behind (either CT scan or MRI) after surgery. MRI will be used during the follow-up period to confirm recurrences from a previous site of DLM.

SUMMARY:
The DREAM study will assess the diagnostic accuracy of diffusion-weighted MRI in combination with other imaging modalities (multiparametric MRI and CT Scan) in determining the true status of disappearing liver metastasis (DLM) detected after conversion systemic therapy for unresectable or borderline resectable colorectal liver metastasis (CRLM).

DETAILED DESCRIPTION:
The advancements of systemic and local therapies for complex CRLM have led to the increased incidence of DLMs. It is hypothesized that DW-MRI imaging could distinguish between a metastasis not completely sterilized by conversion therapy and a sterilized scar (non-viable tumor). If this can be demonstrated, the use of DW-MRI could make a significant impact on the surgical decision making process by providing surgeons a more reliable guide to decide whether to leave behind or to resect/ablate a site of DLM. Most importantly, this surgical choice can also have a significant impact on patient outcomes as it may impact the risk of local recurrence and the need for re-operation.The possibility of improving surgical management of complex CRLM is foreseen if the benefit of observing or resecting small residual metastases and DLMs is clarified through a multi-center and international prospective study.

ELIGIBILITY:
Inclusion Criteria for Eligibility:

1. Contrast-enhanced thorax, abdomen and pelvic CT scan (with at least portal venous phase for the liver) at diagnosis and right before surgery are available
2. Multiparametric MRI at baseline and right before surgery are available (T1/T2, DW-MRI and contrast enhanced MRI).
3. WHO performance status of 0 or 1
4. Previous treatments (chemotherapy, surgery) for primary, liver and extra-hepatic metastases are allowed.
5. No other malignancies in the 3 years prior to study entry with the exception of surgically cured carcinoma in situ of the cervix, in situ breast cancer, incidental finding of stage T1a or T1b prostate cancer gleason score ≤ 6, and basal/squamous cell carcinoma of the skin
6. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the study

Criteria for Enrollment

1. Conversion therapy is either being given or completed
2. Patient is suitable for hepatic resection based on the assessment of MDT composed of at least an expert liver/colorectal surgeon, Gastrointestinal (GI) radiologist and oncologist prior to any liver surgery
3. Hepatic resection is scheduled to take place within 8 weeks of latest imaging

Exclusion Criteria:

1. Contraindications to any contrast agents for CT and MRI or MRI procedure
2. Pregnancy
3. Significant comorbidity that will preclude either conversion therapy or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary tumor histologically proven as colorectal adenocarcinoma, colorectal mucinous adenocarcinoma, colorectal signet ring cell carcinoma or colorectal adenosquamous carcinoma
  Unresectable or borderline resectable liver metastases at the time of diagnosis for liver metastases. Both synchronous and metachronous metastases are allowed
  Age ≥18 years old
  With informed consent
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2016-11; Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Negative Predictive Value (NPV) of the diagnostic imaging (DW-MRI) | 2 years after surgery

SECONDARY OUTCOMES:
NPV of diagnostic imaging among the group of resected confirmed DLMs | 2 years after the surgery
NPV of diagnostic imaging in the group of confirmed DLMs that were left in place | 2 years after ther surgery
NPV of DW-MRI in the group of cDLMs diagnosed by central imaging review | 2 years after the surgery
Correlation between different types of morphologic and ADC changes and TRG to the type of conversion therapy | 2 years after the surgery
Correlation between findings on DW-MRI to histopathology, recurrence rate, complication rates, PFS and OS | 2 years after initial surgery
Long term outcomes of patients who underwent surgery in terms of: - recurrence rates for 2 years after surgery - progression free survival for 2 years after surgery - overall survival for 2 years after surgery | 2 years after initial surgery

CONTACTS AND LOCATIONS:
Overall Officials: Serge Evrard, Study Chair — Institut Bergonie, France
Locations (21):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Innsbruck Universitaetsklinik, Innsbruck, Austria
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Gustave Roussy, Villejuif
- Japan (13):
  - Chiba Cancer Center, Chiba
  - Gifu University Hospital, Gifu
  - Hiroshima Prefectural Hospital, Hiroshima
  - Hyogo College of Medicine, Hyōgo
  - Niigata Prefectural Cancer Center Hospital, Niigata
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - Gunma Cancer Center, Ōta-ku
  - Jichi Medical University Saitama Medical Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - Tokyo Medical and Dental University, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata
  - Kanagawa Cancer Center, Yokohama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kataoka K, Mauer M, Shiozawa M, Marreaud S, Kishi Y, Cabrieto J, Onaya H, Ducreux M, Suto T, Kang HC, Matsuhashi N, Fung A, Yasui M, Rivoire M, Tonooka T, Troisi RI, Nakamura K, Stattner S, Kinugasa Y, Foo WC, Desolneux G, Bonhomme B, Ikeda M, Caballero C, Lordick F, Kanemitsu Y, Evrard S. Diagnostic Accuracy of Imaging in Assessing Nonviability of Disappearing Colorectal Liver Metastasis. JAMA Surg. 2025 Nov 1;160(11):1212-1220. doi: 10.1001/jamasurg.2025.3600. PMID 40960802